CLINICAL TRIAL: NCT01077843
Title: A Nested Case-control Post-authorization Safety Study of Etoricoxib and Other Anti-inflammatory Therapies in a Cohort of Patients With Ankylosing Spondylitis (AS) in the UK, France and Germany
Brief Title: Post-authorization Safety Study of Etoricoxib and Other Anti-inflammatory Therapies in European Patients With Ankylosing Spondylitis (MK-0663-163)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0663-163
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etoricoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure: Ankylosing spondylitis patients currently exposed to anti-inflammatory treatments
  Interventions: Drug: Etoricoxib; Drug: Other Cox-2 inhibitors; Drug: Other Non-selective NSAIDs
- Non-exposure: Ankylosing spondylitis patients not currently exposed to anti-inflammatory treatments
  Interventions: Other: No anti-inflammatory treatment

INTERVENTIONS:
Drug: Etoricoxib — Cox-2 inhibitor
  Other Names: ARCOXIA®
  Groups: Exposure
Drug: Other Cox-2 inhibitors — Cox-2 inhibitor
  Groups: Exposure
Drug: Other Non-selective NSAIDs — Non-selective NSAID
  Groups: Exposure
Other: No anti-inflammatory treatment — No anti-inflammatory prescription
  Groups: Non-exposure

SUMMARY:
This study is a population-based cohort of patients with ankylosing spondylitis (AS) from general medical practices in the UK, France, and Germany with a nested case control component to assess associations between drug exposures of interest and clinical outcomes relevant to patients using cyclooxygenase-2 (COX-2) inhibitors / nonsteroidal anti-inflammatory drugs (NSAIDS).

The main objective of the study is to describe in European participants with AS: 1) the use of etoricoxib 2) characteristics of those who use etoricoxib. 3) the safety profile of etoricoxib and other anti-inflammatory therapies with respect to specific clinical outcomes of interest relative to non-use of these medications and relative to each other.

ELIGIBILITY:
Inclusion Criteria:

* A recorded Ankylosing Spondylitis diagnosis in the database
* A recorded AS diagnosis following the applicable "acceptable data quality" date for the database that contains the patient's records
* At least 6 months of registered medical records in the database after the applicable "acceptable data quality" date as described above, and prior to the recorded AS diagnosis
* Complete information on gender and birth year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will use the combination of the General Practice Research Database (GPRD) in the UK, The Health Improvement Network (THIN) database in the UK, and the IMS Disease Analyzer Database (Disease Analyzer) in the UK, France and Germany.
Sampling Method: Non-Probability Sample
Enrollment: 27381 (Actual)
Dates: Start 2009-08-17 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of gastrointestinal ulcer, perforation or bleeding | First incident event for a given patient through 31-December-2017
Incidence rate of fatal or non-fatal acute myocardial infarction or unstable angina pectoris | First incident event for a given patient through 31-December-2017
Incidence rate of fatal or non-fatal ischemic stroke, or transient ischemic attack | First incident event for a given patient through 31-December-2017
Incidence rate of fatal or non-fatal hemorrhagic stroke | First incident event for a given patient through 31-December-2017
Incidence rate of deep venous thrombosis, pulmonary embolism, or peripheral arterial embolism or thrombosis | First incident event for a given patient through 31-December-2017
Incidence rate of acute renal impairment or failure | First incident event for a given patient through 31-December-2017
Incidence rate of hypertension | First incident event for a given patient through 31-December-2017
Incidence rate of congestive heart failure or left ventricular dysfunction | First incident event for a given patient through 31-December-2017
Incidence rate of sudden or unexplained death | First incident event for a given patient through 31-December-2017

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- See also: EU PAS Register (EUPAS19094) — http://www.encepp.eu/encepp/viewResource.htm?id=19095